CLINICAL TRIAL: NCT03188913
Title: Major Burns Coagulation and the Role of Factor XIII: A Descriptive Study
Brief Title: Factor XIII in Major Burns Coagulation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(ATR)341/2016
Record Dates: First submitted 2017-05-31; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Burns; Coagulation Disorder; Factor XIII Deficiency; Cicatrization; Endothelial Dysfunction
Keywords: Burns; Coagulation; Factor XIII; Glycocalix; Cicatrization
MeSH Terms: conditions — Burns; Hemostatic Disorders; Factor XIII Deficiency; Cicatrix; Thrombosis | interventions — Blood Coagulation Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coagulation tests — The following plasma values will be measured: prothrombin time, activated partial thromboplastin time, thrombin time, functional fibrinogen, lactate, base excess, fibrin monomers, Factor XIII, Factor XII, Factor VIII, Fact von Willebrand, Plasmin, Plasminogen, Alpha-2-antiplasmin, antithrombin, protein C, Heparan sulfate, synecan 1. Surveys on the state of healing and moisture titration will be performed using Tewamether
  Other Names: Cicatrization tests

SUMMARY:
Prospective observational study in which FXIII levels and coagulation tests and cicatrization are measured during the 30 days after the thermal trauma.

DETAILED DESCRIPTION:
This is a prospective observational pilot study in which the levels of FXIII and coagulation, anticoagulation, fibrinolysis, endothelial tissue damage and cicatrization are at the arrival of the patient to hospital, 24 hours before the first surgical intervention, 24h After the first surgical intervention, at 7 days after the first intervention and at 30 days after the thermal trauma, in this moment the healing will also be evaluated. All burn patients who meet the proposed inclusion criteria will be included and entered into the Burn Unit of the Vall d'Hebron University Hospital from the start of the study until reaching a minimum of 20 cases or a temporary term of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Burned patients with a burned body surface of 20% or more
* Over 18 years of age

Exclusion Criteria:

* ABSI (Abbreviated Burns Severity Index) greater than or equal to 12
* Associated polytrauma
* Coagulation deficit previously known
* Treatment with anticoagulants
* Electrocution burns
* Admission into the unit after hour 6 after thermal trauma
* The refusal of the patient, familiar or responsible to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Burned patients over 18 years of age with a burned body surface of 20% or more admitted to the burn unit of the Vall d'Hebron University Hospital from the start of the study to the end of the study with surgical burns ( Second grade or third grade) and for whom informed consent has been obtained
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-19 (Estimated); Primary Completion 2019-06-19 (Estimated); Study Completion 2019-07-21 (Estimated)

PRIMARY OUTCOMES:
Factor XIII | 30 days
  Blood Coagulation Factor XIII levels

SECONDARY OUTCOMES:
Prothrombin Time (PT) | 30 days
  Prothrombin Time blood levels
Activated Partial Thromboplastin Time (APTT) | 30 days
  Activated Partial Thromboplastin Time blood levels
Thrombin Time (TT) | 30 days
  Thrombin Time blood levels
Fibrinogen | 30 days
  Functional fibrinogen blood levels
Lactate | 30 days
  Lactate blood levels
Base Excess (BE) | 30 days
  Base Excess blood levels
Fibrin monomers | 30 days
  Fibrin monomers blood levels
Factor XII | 30 days
  Factor XII blood levels
Factor VIII | 30 days
  Factor VIII blood levels
Factor von Willebrand | 30 days
  Factor von Willebrand blood levels
Plasmin | 30 days
  Plasmin blood levels
Plasminogen | 30 days
  Plasminogen blood levels
Alpha-2-antiplasmin | 30 days
  Alpha-2-antiplasmin blood levels
Antithrombin (AT) | 30 days
  Antithrombin blood levels
Protein C | 30 days
  Protein C blood levels
Heparan sulfate | 30 days
  Heparan sulfate blood levels
Syndecan 1 | 30 days
  Syndecan 1 blood levels
Healing Vancouver test | 30 days
  The Vancouver survey will be conducted on the state of healing
Healing POSAS test | 30 days
  The POSAS survey will be conducted on the state of healing
Tewamether moisture titration | 30 days
  Tewamether consists of two pairs of sensors to measure the humidity and temperature gradients in two different spacings
Surgical bleeding survey | 10 days
  A surgical team survey will be performed on intraoperative bleeding (during the first debridal surgery)
Reintervention due to bleeding | 11 days
  The need of reintervention because of bleeding within the next 24 hours after the first debridal surgery will be registered
Surface debrided | 10 days
  The percentage of debrided surface and type of debridement (in the first debriding surgery)
Surgery Bleeding | 15 days
  Estimated bleeding according to the modified Gross formula (in the first debriding surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Guilabert, MD, Principal Investigator — Vall d'Hebron Universitary Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guilabert P, Usua G, Martin N, Abarca L, Barret JP, Colomina MJ. Fluid resuscitation management in patients with burns: update. Br J Anaesth. 2016 Sep;117(3):284-96. doi: 10.1093/bja/aew266. PMID 27543523
- [Background] Glas GJ, Levi M, Schultz MJ. Coagulopathy and its management in patients with severe burns. J Thromb Haemost. 2016 May;14(5):865-74. doi: 10.1111/jth.13283. Epub 2016 Mar 23. PMID 26854881
- [Background] Sherren PB, Hussey J, Martin R, Kundishora T, Parker M, Emerson B. Lethal triad in severe burns. Burns. 2014 Dec;40(8):1492-6. doi: 10.1016/j.burns.2014.04.011. Epub 2014 Jul 1. PMID 24996247
- [Background] Sherren PB, Hussey J, Martin R, Kundishora T, Parker M, Emerson B. Acute burn induced coagulopathy. Burns. 2013 Sep;39(6):1157-61. doi: 10.1016/j.burns.2013.02.010. Epub 2013 Mar 14. PMID 23498713
- [Background] King DR, Namias N, Andrews DM. Coagulation abnormalities following thermal injury. Blood Coagul Fibrinolysis. 2010 Oct;21(7):666-9. doi: 10.1097/MBC.0b013e32833ceb08. PMID 20689402
- [Background] Mitra B, Wasiak J, Cameron PA, O'Reilly G, Dobson H, Cleland H. Early coagulopathy of major burns. Injury. 2013 Jan;44(1):40-3. doi: 10.1016/j.injury.2012.05.010. Epub 2012 Jun 5. PMID 22677221
- [Background] Lavrentieva A, Kontakiotis T, Bitzani M, Papaioannou-Gaki G, Parlapani A, Thomareis O, Tsotsolis N, Giala MA. Early coagulation disorders after severe burn injury: impact on mortality. Intensive Care Med. 2008 Apr;34(4):700-6. doi: 10.1007/s00134-007-0976-5. Epub 2008 Jan 12. PMID 18193192
- [Background] Barret JP, Dziewulski PG. Complications of the hypercoagulable status in burn injury. Burns. 2006 Dec;32(8):1005-8. doi: 10.1016/j.burns.2006.02.018. Epub 2006 Aug 1. PMID 16879922
- [Background] Barret JP, Gomez PA. Disseminated intravascular coagulation: a rare entity in burn injury. Burns. 2005 May;31(3):354-7. doi: 10.1016/j.burns.2004.11.006. Epub 2005 Jan 21. PMID 15774294
- [Background] Aoki K, Aikawa N, Sekine K, Yamazaki M, Mimura T, Urano T, Takada A. Elevation of plasma free PAI-1 levels as an integrated endothelial response to severe burns. Burns. 2001 Sep;27(6):569-75. doi: 10.1016/s0305-4179(01)00011-0. PMID 11525850
- [Background] Levin GY, Egorihina MN. The role of fibrinogen in aggregation of platelets in burn injury. Burns. 2010 Sep;36(6):806-10. doi: 10.1016/j.burns.2009.05.005. Epub 2010 Mar 16. PMID 20236770
- [Background] Schaden E, Hoerburger D, Hacker S, Kraincuk P, Baron DM, Kozek-Langenecker S. Fibrinogen function after severe burn injury. Burns. 2012 Feb;38(1):77-82. doi: 10.1016/j.burns.2010.12.004. Epub 2011 Nov 23. PMID 22113102
- [Background] Nielsen VG, Gurley WQ Jr, Burch TM. The impact of factor XIII on coagulation kinetics and clot strength determined by thrombelastography. Anesth Analg. 2004 Jul;99(1):120-123. doi: 10.1213/01.ANE.0000123012.24871.62. PMID 15281516
- [Background] Korte W. [Fibrin monomer and factor XIII: a new concept for unexplained intraoperative coagulopathy]. Hamostaseologie. 2006 Aug;26(3 Suppl 1):S30-5. German. PMID 16953290
- [Background] Jambor C, Reul V, Schnider TW, Degiacomi P, Metzner H, Korte WC. In vitro inhibition of factor XIII retards clot formation, reduces clot firmness, and increases fibrinolytic effects in whole blood. Anesth Analg. 2009 Oct;109(4):1023-8. doi: 10.1213/ANE.0b013e3181b5a263. PMID 19762725